CLINICAL TRIAL: NCT03585738
Title: Effects of Oral Inositol Supplementation on Obstetrics Outcomes in Polycystic Ovary Syndrome Women After Spontaneous Conception
Brief Title: Effects of Oral Inositol Supplementation on Obstetrics Outcomes in PCOS Women
Acronym: IPOSI-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPOSI-1
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Inositol; Polycystic ovarian syndrome; Pregnancy; Obstetrics outcomes; Gestational diabetes; Preeclampsia
MeSH Terms: conditions — Polycystic Ovary Syndrome; Diabetes, Gestational; Pre-Eclampsia | interventions — Inositol; Folic Acid

STUDY DESIGN:
Intervention Model Description: Randomized multi centre double-blind controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, care provides, investigators and outcome assessors are blinded for the treatment: Inositol + Folic acid versus Folic acid alone. The treatment allocation is identified by code number before the study start, and will be revealed only after data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inositol + Folic acid (Experimental): Couples with PCOS infertile women, diagnosed according to the Rotterdam criteria, who access infertility center with conception desire. These women will receive oral supplementation with Inositol (Myo-inositol and D-chiro-inositol at 40:1 ratio) plus Folic acid before spontaneous conception until delivery.
  Interventions: Dietary Supplement: Inositol + Folic acid
- Folic acid (Placebo Comparator): Couples with PCOS infertile women, diagnosed according to the Rotterdam criteria, who access infertility center with conception desire. These women will receive oral supplementation with Folic acid before spontaneous conception until delivery.
  Interventions: Dietary Supplement: Folic acid

INTERVENTIONS:
Dietary Supplement: Inositol + Folic acid — Daily oral supplementation before spontaneous conception until delivery:
  Myo-Inositol: 1100 mg D-chiro-inositol: 27.6 mg Folic acid: 400 mcg
  Arms: Inositol + Folic acid
Dietary Supplement: Folic acid — Daily oral supplementation before spontaneous conception until delivery:
  Folic acid: 400 mcg
  Arms: Folic acid

SUMMARY:
Polycystic ovarian syndrome (PCOS) is a heterogeneous, multifaceted and complex disorder characterized by insulin resistance (IR), hyperinsulinemia, and hyperandrogenism leading ovarian disfunction and infertility. Given the central pathogenic role of IR in the endocrine, reproductive, and metabolic disturbances of PCOS, several pharmacological and non-pharmacological approaches have been proposed to counteract the hyper insulinemic IR typical of the syndrome. Two Inositol stereoisomers, Myo-Inositol (MI) and D-chiro-inositol (DCI), captured the attention of researchers for their insulin-sensitizing actions, which configure them as proper candidates for the treatment of PCOS.

Very few studies reported on spontaneous clinical pregnancy rates, none were powered for this outcome, and none reported on the clinically relevant outcome of live birth. Therefore, data about clinical pregnancy rate, live birth rate, and miscarriage rate comparing inositols with placebo are limited.

Nevertheless, regarding infertility the primary outcomes that should be considered are clinical pregnancy rate, miscarriage rate and live birth rate. Although many studies showed improved hormonal and metabolic profile and improved ovulation rate and higher quality and number of oocyte retrieved in Assisted Reproductive Technology (ART) in PCOS women after inositols administration, data about clinical pregnancy rate, live birth rate, and miscarriage rate are limited with several concerns regarding interpretation of the studies.

Furthermore, independently by the effect on PCOS related infertility, few data are available about the role of inositol on obstetrics outcomes of pregnancies conceived after treatment with inositol and/or orally supplemented during pregnancy. Considering that the combination of MI and DCI alleviate many of the metabolic dysregulations typical of PCOS thanks to insulin-sensitizing actions, it is plausible consider a beneficial effects on pregnancy complications such as gestational diabetes and preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy spontaneously conceived in women with PCOS diagnosed by Rotterdam criteria that starts oral supplementation before conception.

Exclusion Criteria:

* Any kwon pre-pregnancy disease.
* Any other pharmacological, non-pharmacological or nutraceutical treatment (beside oral folic acid supplementation) more than 3 months before the enrollment (wash-out period) or during the trial, or until the development or pregnancy-induced/related diseases requiring pharmacological treatments.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes prevalence | During pregnancy at 16-18 week or 24-28 weeks as recommended
  Gestational diabetes prevalence: number of women that develop gestational diabetes diagnosed based on oral glucose tolerance test (OGTT) cut-off (92 - 180 - 153 mg/dl).
Preeclampsia prevalence | During pregnancy after the 20 week of gestation
  Preeclampsia prevalence: number of women that develop preeclampsia diagnosed based on blood pressure higher than 140/90 mmHg after 20 week of gestation plus 24h proteinuria higher that 300mg.
Birth weight | At delivery.
  gr
Weight gain in pregnancy | Change in weight before pregnancy and at the 38 week of gestation
  Kg

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Simone Garzon, M.D., Principal Investigator — Univerisity of Verona; Fabio Ghezzi, M.D., Study Chair — Università degli Studi dell'Insubria; Massimo Franchi, M.D., Study Chair — Univerisity of Verona; Antonella Cromi, M.D., Principal Investigator — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided